CLINICAL TRIAL: NCT00000582
Title: Cooperative Study of Factor VIII Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: 302
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Blood Coagulation Disorders; Hematologic Diseases; Hemophilia A; Hemorrhagic Disorders
MeSH Terms: conditions — Blood Coagulation Disorders; Hematologic Diseases; Hemophilia A; Hemorrhagic Disorders | interventions — Factor IX

INTERVENTIONS:
Drug: factor ix

SUMMARY:
To test the efficacy of prothrombin complex concentrates (Factor IX) in the treatment of hemophiliac patients who had inhibitors to Factor VIII.

DETAILED DESCRIPTION:
BACKGROUND:

Despite major advances in the treatment of patients with hemophilia, a serious remaining challenge was presented by the occurrence of circulating inhibitors to Factor VIII. Because of lack of information on the natural course of patients with Factor VIII inhibitors, the relative efficacy of various modes of therapy was not established. The Division of Blood Diseases and Resources decided to sponsor a clinical investigation which would evaluate populations of hemophilia patients for Factor VIII inhibitors, follow up these patients to provide information on the natural history of the inhibitor in the hemophilia patients, and make available a reference center to monitor results and attain uniformity.

Treatment of a patient with a severe inhibitor and consequent bleeding remained a problem. Management included protracted treatment with Factor VIII, use of immunosuppressive agents and prothrombin complex (or Factor IX) concentrates. The rationale for Factor IX was that it bypassed the defect in Factor VIII caused by the inhibitor. This method of therapy attracted wide popularity, but the success was greatly debated. It was intended at the very outset of the Factor VIII study that therapeutic trials involving patients with inhibitors would not be a prime function, but that such studies would be monitored if necessary. A controlled trial of Factor IX concentrates therapy was strongly advised by the DBDR Advisory Committee. Accordingly, during fiscal year 1978, a protocol for a double-blind control study was developed by the Factor VIII inhibitor group. The trial began in the spring of 1978, and the intervention terminated about one year later.

DESIGN NARRATIVE:

Double-blind study; patients served as their own controls. A total of 51 patients each received a single large dose of Konyne, Proplex, or diluted albumin (as a control). Joint bleeding of the elbow, knee, and ankle was evaluated six hours after each dose.

ELIGIBILITY:
Males with hemophilia, not stratified as to ethnic group.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1978-07; Study Completion 1979-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Aledort — Icahn School of Medicine at Mount Sinai; J. Edson — University of Minnesota; M. Eyster — Milton S. Hershey Medical Center; Scott Goodnight — University of Oregon Health Sciences Center; William Hathaway — University of Colorado Medical Center; Jack Lazerson — Milwaukee Children's Hospital; Peter Levine — Memorial hospital; Jeanne Lusher — Wayne State University; Campbell McMillan — University of North Carolina; Sandor Shapiro — Thomas Jefferson University

REFERENCES:
- [Background] Eyster ME, Gill FM, Blatt PM, Hilgartner MW, Ballard JO, Kinney TR. Central nervous system bleeding in hemophiliacs. Blood. 1978 Jun;51(6):1179-88. No abstract available. PMID 647123
- [Background] Lusher JM, McMillan CW. Severe factor VIII and factor IX deficiency in females. Am J Med. 1978 Oct;65(4):637-48. doi: 10.1016/0002-9343(78)90852-5. PMID 309282
- [Background] Kasper CK. Effect of prothrombin complex concentrates on factor VIII inhibitor levels. Blood. 1979 Dec;54(6):1358-68. PMID 508942
- [Background] Lusher JM, Shapiro SS, Palascak JE, Rao AV, Levine PH, Blatt PM. Efficacy of prothrombin-complex concentrates in hemophiliacs with antibodies to factor VIII: a multicenter therapeutic trial. N Engl J Med. 1980 Aug 21;303(8):421-5. doi: 10.1056/NEJM198008213030803. PMID 6771653
- [Background] Gerety RJ, Eyster ME, Tabor E, Drucker JA, Lusch CJ, Prager D, Rice SA, Bowman HS. Hepatitis B virus, hepatitis A virus and persistently elevated aminotransferases in hemophiliacs. J Med Virol. 1980;6(2):111-8. doi: 10.1002/jmv.1890060203. PMID 6264019